CLINICAL TRIAL: NCT06816979
Title: Assessing the CSF-ctDNA of Patients With Stage III and IV Non-Small Cell Lung Cancer: A Pilot Study
Brief Title: Lumbar Punctures for the Detection of ctDNA in the Cerebrospinal Fluid of Patients With Stage III and IV Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Joshua Palmer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-22032; NCI-2023-03242 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-11-04; First posted 2025-02-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Spinal Puncture; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1: Stage III/IV without brain metastases (LP) (Experimental): Patients undergo LP for collection of CSF and blood sample collection after completion of chemoradiotherapy (stage III) or after diagnosis (stage IV) on study. Patients also undergo MRI during screening and 12 month follow-up.
  Patients with CSF negative for ctDNA at the first LP draw, undergo an additional LP draw at 6 months. Patients with CSF positive for ctDNA at the first LP draw, may not undergo an additional LP at 6 months.
  Interventions: Procedure: Biospecimen Collection; Procedure: Lumbar Puncture; Device: Magnetic Resonance Imaging
- Cohort 2: Stage IV NSCLC with brain metastases (LP) (Experimental): Patients undergo LP for collection of CSF and blood sample collection on study. Patients also undergo MRI during screening.
  Patients with CSF negative for ctDNA at the first LP draw, undergo an additional LP draw at 6 months. Patients with CSF positive for ctDNA at the first LP draw, may not undergo an additional LP at 6 months.
  Interventions: Procedure: Biospecimen Collection; Procedure: Lumbar Puncture; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Device: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase I trial assesses the use of lumbar punctures to detect whether there is circulating tumor deoxyribonucleic acid (ctDNA) in the fluid that surrounds the brain and spinal cord (cerebrospinal fluid) in patients with stage III and IV non-small cell lung cancer (NSCLC). Patients with stage III and IV NSCLC are at risk of having their cancer spread from where it first started to the brain (metastatic). Because of this, more effective prognostic tools are necessary to determine which stage III and IV NSCLC patients are more likely to develop brain metastases. Cerebrospinal fluid (CSF) could be a reliable source of ctDNA to confirm and predict the presence of brain metastases in these patients. Assessing cell free DNA shed from tumor cells could be a sensitive and minimally invasive way to detect or characterize metastatic tumors in the central nervous system (CNS). Lumbar puncture is procedure in which a thin needle called a spinal needle is put into the lower part of the spinal column to collect CSF. Lumbar punctures for the collection of CSF may help doctors detect or measure changes in cell types, genes, and proteins of circulating tumor cells related to lung cancer that will help determine the presence of brain metastases which could become a standard of care screening tool utilized in the follow-up of patients diagnosed with stage II or IV NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if CSF-ctDNA positivity in patients with locally advanced lung cancer can predict the presence of brain metastases within a one year period.

II. To prospectively confirm that cerebrospinal fluid (CSF) circulating tumor DNA (ctDNA) can be detected in patients diagnosed with metastatic non-small cell lung cancer (NSCLC) to the brain utilizing next generation sequencing (NGS) and single gene quantitative/biomarker analyses through the CNSide (trademark) platform.

SECONDARY OBJECTIVES:

I. To use the CNSide (trademark) platform to assess for the presence of circulating tumor cells in both CSF and peripheral blood.

II. To compare the NGS profile of the ct-DNA in the CSF with matched peripheral blood samples.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1 (STAGE III/IV NSCLC WITHOUT BRAIN METASTASES): Patients undergo lumbar puncture (LP) for collection of CSF and blood sample collection after completion of chemoradiotherapy (stage III) or after diagnosis (stage IV) on study. Patients also undergo magnetic resonance imaging (MRI) during screening and 12 month follow-up.

COHORT 2 (STAGE IV NSCLC WITH BRAIN METASTASES): Patients undergo LP for collection of CSF and blood sample collection on study. Patients also undergo MRI during screening.

Patients with CSF negative for ctDNA at the first LP draw, undergo an additional LP draw at 6 months. Patients with CSF positive for ctDNA at the first LP draw, may not undergo an additional LP at 6 months.

Patients without brain metastases are followed for 12 months. Patients with brain metastases are followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* New histological diagnosis of stage III or IV NSCLC
* For stage III/IV NSCLC patients without brain metastases, a documented mutation on lung cancer mutation panel (PULMOL) is required
* Patient treated with radiation therapy and/or systemic therapy at Ohio State University
* Estimated survival >= 1 year
* No medical contraindication to lumbar puncture

Exclusion Criteria:

* Patient has Alzheimer's, dementia, or mental disability
* Patient is not able to receive MRI
* Patient has allergy to xylocaine or any numbing medication for lumbar puncture
* Previous cancer history prior to diagnosis of NSCLC
* Pregnant or lactating women, or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the medication and radiation required for standard of care treatment has unknown effects on the unborn fetus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Intracranial disease in locally advanced lung cancer patients | Up to 6 months
  An MRI will be performed six months after lumbar puncture in Cohort One. MRI sequences with T1 post-contrast for disease and structure definition and T2/FLAIR sequences for identification of peri-tumoral edema or cystic volumes will be obtained.
Cerebral spinal fluid- circulating tumor deoxyribonucleic acid (ctDNA) detection rate for lung non-small cell carcinoma patients with metastatic disease to the brain | Up to 12 months
  Will estimate the frequency of ctDNA detection with a 90% Clopper-Pearson confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Palmer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu